CLINICAL TRIAL: NCT03527667
Title: Incentivized Smoking Cessation for Tobacco Treatment-Resistant Diabetics
Brief Title: Incentivized Smoking Cessation for Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Cancer Research UK (Other); University of Strathclyde (Other); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8652
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Smoking Cessation; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Smoking Cessation; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: 3-arm randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short term incentives (Experimental): usual quit smoking treatment (counseling + medication) plus 6-weeks of payments for proof of smoking abstinence
  Interventions: Behavioral: Financial incentives
- Long term incentives (Experimental): usual quit smoking treatment (counseling + medication) plus 12-weeks of payments for proof of smoking abstinence
  Interventions: Behavioral: Financial incentives
- No incentives (No Intervention): usual quit smoking treatment (counseling + medication)

INTERVENTIONS:
Behavioral: Financial incentives — Treatment arm participants will receive financial incentives ($20 per week) contingent on biochemically verified smoking abstinence submitted once daily for the time period allocated.
  Arms: Long term incentives; Short term incentives

SUMMARY:
This pilot study aims to test the feasibility of providing incentives to patients with T2D contingent on remote biochemical verification using a smartphone carbon monoxide (CO) monitor. The investigators will use an ecological momentary assessment (EMA) smartphone application and CO sensor to monitor urges to smoke, stressors, smoking behaviors, and to validate continuous abstinence throughout the intervention. Two different contingency management structures will be explored to investigate the length of time incentives need to be offered.

DETAILED DESCRIPTION:
Individuals with type 2 diabetes (T2D) are at an increased risk of many cancers, though the causal link is not well understood. Continuing to smoke after a T2D diagnosis is also associated with accelerated progression of microvascular and macrovascular complications and an increased risk of death. Smoking cessation is recommended as a standard treatment for diabetes. However, both patients and providers are faced with other challenging lifestyle changes and disease management processes, which lead to greater difficulty in quitting.

Contingency management, or a method of providing financial incentives contingent upon positive behaviors, has shown promise for improving adherence to medication among diabetics and for improving smoking cessation in other populations. This approach could offer an innovative and scalable means of increasing abstinence in this group, ultimately reducing their risk of cancer. This is a multicenter pilot randomized controlled trial that will recruit participants in Oklahoma and in Strathclyde, Scotland.

This pilot study aims to test the feasibility of providing incentives to patients with T2D contingent on remote biochemical verification using a smartphone carbon monoxide (CO) monitor. The investigators will use an ecological momentary assessment (EMA) smartphone application and CO sensor to monitor urges to smoke, stressors, smoking behaviors, and to validate continuous abstinence throughout the intervention. Two different contingency management structures will be explored to investigate the length of time incentives need to be offered. Qualitative semi-structured interviews will be used to explore the patient and provider acceptability of an incentive-based cessation program, any unintended consequences and possible differences between UK and US health settings.

The results of this research will inform the feasibility of carrying out a randomized controlled trial of this intervention. The ultimate aim is to develop an effective intervention that could be scaled to the T2D population at large, which reduces cancer risk and improves disease outcomes among a high-risk group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75
* Type 2 diabetes diagnosis greater than 1 year prior to enrollment
* Currently smoking at least 5 cigarettes per day
* Self-reported quit attempt in past 12 months

Exclusion Criteria:

* Unwilling to make a quit attempt
* Unable to use smartphone iCO monitor following training session

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of CO readings completed | 12 weeks
  Feasibility of study determined by number of CO readings completed by each participant

SECONDARY OUTCOMES:
Quit outcomes | 12 weeks
  Proportion of participants who quit smoking
Cigarettes per day | 12 weeks
  Reduction in cigarettes smoked per day

CONTACTS AND LOCATIONS:
Overall Officials: Sydney A Martinez, PhD, Principal Investigator — University of Oklahoma
Locations (2):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States
- University of Strathclyde, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez SA, Quaife SL, Hasan A, McMillan KA, Beebe LA, Muirhead F. Contingency management for smoking cessation among individuals with type 2 diabetes: protocol for a multi-center randomized controlled feasibility trial. Pilot Feasibility Stud. 2020 Jun 11;6:82. doi: 10.1186/s40814-020-00629-7. eCollection 2020. PMID 32537238